CLINICAL TRIAL: NCT06237088
Title: Mother-infant Connection Strategy Program: Impact on Psychological Distress and Mother-infant Bonding in Women
Brief Title: Mother-infant Connection Strategy Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Wan-Lin Pan, Assistant Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 111-E-21
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Psychological; Mother-Infant Interaction
Keywords: Mindfulness, Anxiety, Depression, Mother-Infant Interaction
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- eight-week mindfulness programs (Active Comparator): The intervention consists of 2.5-hour classes per week over a period of eight weeks.
  Interventions: Other: eight-week mindfulness programs
- online mindfulness program (Experimental): The intervention includes an eight-week internet-based mindfulness program. The program introduces participants to a new mindfulness topic every week. These topics are heavily inspired by the eight-week mindfulness programs.
  Interventions: Other: online mindfulness program
- care as usual (No Intervention): Hospital-based antenatal care involves all aspects of pregnancy, childbirth and postpartum.

INTERVENTIONS:
Other: online mindfulness program — The intervention includes an eight-week internet-based mindfulness program. The program introduces participants to a new mindfulness topic every week. These topics are heavily inspired by the eight-week mindfulness programs.
  Arms: online mindfulness program
Other: eight-week mindfulness programs — The intervention consists of 2.5-hour classes per week over a period of eight weeks.
  Arms: eight-week mindfulness programs

SUMMARY:
This study evaluated the long-term effects of an online mindfulness-based program on the psychological distress and mother-infant bonding of women

DETAILED DESCRIPTION:
The aim of this study was to test the efficacy of an online mindfulness program in reducing women's perceived stress, anxiety, depression, and in enhancing mindfulness and mother-infant bonding compared to a control group. The investigators hypothesize that the use of an online mindfulness program or an eight-week mindfulness program by the two experimental groups will lead to improved mood symptoms and mother-infant bonding compared with the control group.

A randomized controlled trial comparing three groups of healthy, singleton pregnant women was conducted using the Random Allocation Software (Saghaei, 2004). We used G-Power 3.1.9 for Windows to analyze the minimum effect size that would be statistically significant with an 80% probability, using an alpha error probability of 0.05 in the "ANOVA: Repeated measures, between factors" option. We inputted 3 for the number of groups, 4 for the number of measurements, 0.5 for the correlation between repeated measures, and factored in a 20% attrition rate. There are 41 women in each group.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were at the age over 18
* Could speak and read Chinese fluently
* Willing and be ale to attend the education program

Exclusion Criteria:

* Taking medication for diagnosing mental illness
* With complicated or high-risk pregnancies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
anxiety | baseline , and at eight weeks (after the intervention), 36 weeks of gestation, and the follow-up at 2 , 4 months postpartum
  The Beck Anxiety Inventory using 21 items on the scale describes a symptom of anxiety. Responses are rated from 0 (never) to 3 (very often), with higher scores corresponding to higher perceived anxiety.
depression | baseline , and at eight weeks (after the intervention), 36 weeks of gestation, and the follow-up at 2 , 4 months postpartum
  Edinburgh Perinatal Depression Scale, that was 10-question questionnaire provides a valuable and efficient way to identify patients at risk of perinatal depression. Each item is scored from 0 to 3, with item scores summed to produce a total score
mindfulness | baseline , and at eight weeks (after the intervention), 36 weeks of gestation, and the follow-up at 2 , 4 months postpartum
  The Five Facet Mindfulness Questionnaire, that was 39-item is based on factor analysis. The five facets of the FFMQ include: observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience. Scoring uses a 5-point Likert scale, with 1 representing "never or very rarely true" and 5 representing "very often or always true"
mother-infant bonding | the follow-up at 2 , 4 months postpartum.
  The Postpartum Bonding Questionnaire, that was 25 items, with four factors. The first factor was labelled general emotional factor, the second anger towards and rejection of baby; the third infant-focus anxiety; and the fourth, risk of abuse.

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Lin Pan, PHD, Principal Investigator — assistant professor
Locations (1):
- Wan-Lin Pan, Taipei, Taiwan